CLINICAL TRIAL: NCT07276451
Title: Effectiveness of the Digital Mental Health Intervention and Open Peer Support Platform in Improving Participant Quality of Life: a Randomised Controlled Trial.
Brief Title: Effectiveness of the DMHI and OPS Platform in Improving Participant QOL: a Randomised Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Dmitry Shamenkov, Dr., Universidade Nova de Lisboa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21/2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Depression and Quality of Life; Quality of Life
Keywords: digital mental health intervention; open peer support; mental health; online support
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention group will immediately be granted 30 days of access to the Platform and its resources (see 3.4.). The control group will be granted access to the Platform following a second round of assessment on day 31. The intervention group will also be required to complete outgoing assessment on day 31.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers responsible for participant enrolment and data collection remain blinded to the randomization sequence until after the completion of the study. Allocation concealment is maintained by securely storing the randomization sequence and ensuring that access is restricted to an authorised expert. Only the authorised expert will participate in generating random allocation and securing the data until the intervention phase is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Intervention group) (Experimental): Intervention group. Participants in the intervention group will be analysed according to their QOL scores and feedback on secondary conditions will be used for pooling and subgroup analyses. Participant in the intervention group will be determined through a randomised selection.
  Interventions: Other: Participation in digital mental health intervention and open peer support platform
- Group 2 (control group) (No Intervention): Participants in the control group, included as a result of randomised selection, will be put on the waitlist to access the Platform throughout the duration of the trial. The control group participants will be granted access to the Platform on day 31 of the trial. The introductory and closing evaluations will be performed on both groups at similar time points. This group is the waitlist group.

INTERVENTIONS:
Other: Participation in digital mental health intervention and open peer support platform — Participants in the experimental group will be immediately enrolled in the Platform and will have access to several interactive (daily mindfulness exercises; open dialogue group sessions; peer support forum; mentor chat) and passive (resource library: pre-recorded videos and guides) components for a total of 30 days, after which a final assessment will be performed on day 31. Control group participants will not be granted access to the Platform through the duration of the trial.
  Arms: Group 1 (Intervention group)

SUMMARY:
RCT to evaluate the efficacy of a digital mental health intervention platform with open peer support in improving participant quality of life.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the role of the DHMI and OPS platform (further referred to as "the Platform") in improving participants' QOL. Participants will be recruited through community outreach, advertisements in healthcare facilities, and online platforms (See Appendix 2 for sample advertisements and Appendix 5 for list of centres for potential outreach). The RCT will be a parallel study where participants are randomly assigned to one of the groups using computer-generated random allocation. Prior to enrolment, participants will be assessed on eligibility and given initial assessment scales to evaluate their mental, physical states, the results of which will be reviewed by study supervisors and a local clinical specialist, who will perform risk assessment and when needed recommend exclusion and referral to specialized care facilities, based on participant scores. Upon enrolment, the participants will be randomly assigned to one of two groups: intervention group and control group. The intervention group will immediately be granted 30 days of access to the Platform and its resources. The control group will be granted access to the Platform following a second round of assessment on day 31. The intervention group will also be required to complete outgoing assessment on day 31.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* No current clinical diagnosis of a mental health disorder;
* No mental-health treatment or psychotropic medication initiated within the past 3 months;
* Able to access the internet and provide informed consent.

Exclusion Criteria:

* Current engagement with a mental health professional or therapy;
* Inability to access the DMHI and OPS platform, or inability to provide informed consent;
* PHQ-9 score ≥15 or GAD-7 score ≥15 at baseline (these participants will be referred to specialist services and excluded from further study participation)

Confirmation of eligibility to participate. To comply with local regulations and ensure participant safety, a qualified and appropriately licensed specialist, affiliated with the institution will participate in screening of the participants recruitment results and carrying out decisions on whether to include or exclude the participant from the study based on degree of severity in the underlying psychological or psychiatric condition. The decision to exclude participants will be made based on safety considerations, need for emergency psychiatric help, compliance assumption and perceived efficacy.

Withdrawal. Participation is voluntary. All enrolled participants are free to withdraw from the study at any time with or without notice to study personnel.

Risk to self and/or others. During enrollment and study course, participants will be screened for severity of symptoms. If our participating specialist identifies a risk to self or others, appropriate actions will be taken to contact the authorities and local law representatives according to European and Local Law.

Sample size estimates. For two groups and a dichotomous endpoint (improvement or no improvement) and an anticipated incidence of 45% in the intervention group and 75% in the control group, at a 95% confidence level and 5% margin of error, power of 80% and enrolment ratio of 1, a sample size of 82 participants was chosen for this RCT (41 in intervention group, 41 in control group).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome (WHOQOL-BREF change 0-31) | 1 month
  Change in Overall Quality of Life, as measured by the WHOQOL-BREF total score, from baseline (day 0) to post-intervention (day 31), treated as a continuous variable. A clinically meaningful improvement is defined a priori as a ≥10% increase from baseline.

SECONDARY OUTCOMES:
SWLS | 1 month
  Satisfaction with life assessed using measures such as the Satisfaction with Life Scale (SWLS).
PSS | 1 month
  Stress levels assessed using the Perceived Stress Scale (PSS).
GAD-7 | 1 month
  Anxiety levels measured using the Generalised Anxiety Disorder 7-item Scale (GAD-7).
PHQ-9 | 1 month
  Depression severity evaluated using the Patient Health Questionnaire 9-item (PHQ-9)
Social Connectedness | 1 month
  Communitas Scale for assessing social connectedness
MLQ | 1 month
  Meaning of Life Questionnaire (MLQ).

OTHER OUTCOMES:
Mediator: adherence to platform | 1 month
  Adherence to platform (measured by rate of interaction)
Mediator: concomitant medication use | 1 month
  Concomitant medication use.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided